CLINICAL TRIAL: NCT05722028
Title: Predictive Factors for Successful Operative Hysteroscopy Using Tissue Removal Device (TruClear System) Without Anesthesia
Status: Completed | Type: Observational
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Principal Investigator, Maayan Gal, investigator, Assaf-Harofeh Medical Center
Other Study IDs: 123456
Record Dates: First submitted 2023-01-29; First posted 2023-02-10 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Uterine Polyp; Retained Products of Conception
MeSH Terms: interventions — Hysteroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Patients with benign uterine findings (polyp / retained products of conception): Female patients undergoing diagnostic hysteroscopy with a diagnosis of uterine polyp or retained products of conception. These patients are then invited to a surgical office procedure without anaesthesia to remove these findings.
  Interventions: Procedure: hysteroscopy

INTERVENTIONS:
Procedure: hysteroscopy — Surgical hysteroscopy without anaesthesia for removal of uterine polyp / retained products of conception.

SUMMARY:
Background: Small-diameter operative hysteroscopes may allow to perform operative hysteroscopy without general anesthesia in selected patients. One of these instruments is the tissue removal device (TRD), which resects and removes intrauterine pathology such as endometrial polyps and retained products of conception (RPOC) with a diameter of ¬6 mm.

Objective: To assess the success rate and intraoperative pain of patients undergoing operative hysteroscopy without anesthesia with the TRD (TruClear Elite Mini-Hysteroscope) for removal of endometrial polyps or RPOC.

Methods: Prospective observational study. Participation in the study was offered to patients diagnosed with uterine polyps or RPOC on office diagnostic hysteroscopy. The patients filled out a digital questionnaire before and after the operation. A successful procedure was defined as complete hysteroscopic removal of the uterine pathology using the TruClear system. Oral 400 mcg misoprostol 12 hours before the procedure was prescribed for cervical ripening.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of polyp or retained products of conception in diagnostic hysteroscopy.
* Medical need to remove the finding according to accepted criteria.
* Patient's consent to the removal of the finding in a procedure without anesthesia.
* Patient's consent to participate in the study.

Exclusion Criteria:

* Any indication for performing the procedure under anesthesia in an operating room, such as:

  1. Medical background requiring operation in an operating room.
  2. Personal / mental background requiring procedure under general anesthesia.
  3. Cervical stenosis
  4. Previous failure to remove the finding in a procedure without anesthesia
  5. Lack of response to performing the operation without anesthesia
* The lack of response to participate in the study
* A known diagnosis of malignancy from a previous sample of the polyp or endometrium

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Women who have been diagnosed with a benign pathology (polyp or retained products of conception) in diagnostic hysteroscopy and are accepted for surgical hysteroscopy in a clinical setting (without anesthesia) for its removal.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Procedure completed successfully | Immediately after procedure
  Was the procedure completed - yes/no

SECONDARY OUTCOMES:
Prevalence of VAS (pain scale) > 5 during procedure | Immediately after procedure
  VAS (Visual analogue scale 0-10, most painful 10) grading by the patient
Prevalence of VAS (pain scale) > 5, five minutes after procedure | 5 minutes after procedure
  VAS (Visual analogue scale 0-10, most painful 10) grading by the patient
Acceptable procedure by the patient | 5 minutes after procedure
  Was the procedure acceptable by the patient (1-4 when 1 is most acceptable)
Recommended procedure by the patient | 5 minutes after procedure
  Would the patient recommend her acquittance the procedure in this outline (1-5, most recommended 5) aquitance (1-5)

CONTACTS AND LOCATIONS:
Locations (1):
- Shamir medical center, Zrifin, Israel